CLINICAL TRIAL: NCT05474456
Title: Effects of Sustained Natural Apophyseal Glides Versus Cervical Manipulation on Pain and Disability in Non Specific Neck Among Wrestlers
Brief Title: Effects of Sustained Natural Apophyseal Glides Versus Cervical Manipulation on Pain and Disability in Wrestle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0403
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Neck Pain; Disability Physical
Keywords: Pain; Neck Injury; Snags; Cervical Manipulation; Disability
MeSH Terms: conditions — Neck Pain; Pain; Neck Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNAGs Group (Experimental): Group A sustained natural apophyseal glides will be provided to wrestlers in the sitting position. SNAG technique applied on the dorsal side of the neck. The treatment will be given for 6 weeks, 2 sessions per week.
  Interventions: Other: SNAGs
- Manipulation Group (Active Comparator): group bWrestlers will be treated with high velocity, low amplitude thrust. The treatment will be given for 6 weeks, 2 sessions per week.
  Interventions: Other: Manipulation

INTERVENTIONS:
Other: SNAGs — Wrestlers will be treated with high velocity, low amplitude thrust. The treatment will be given for 6 weeks, 2 sessions per week.
  Arms: SNAGs Group
Other: Manipulation — Wrestlers will be treated with high velocity, low amplitude thrust. The treatment will be given for 6 weeks, 2 sessions per week.
  Arms: Manipulation Group

SUMMARY:
This study will be conducted to evaluate effect of sustained natural apophyseal glides and cervical manipulation in pain and disability of neck among wrestler players .All subjects will be selected between ages 18 to 35 years. Data will be collected from players in registered gujranwala wrestling clubs. Study design will be Randomized Clinical Trial. Neck pain disability index questionnaire and NPRS will be used to check the disability in neck and intensity of pain respectively. Informed consent will be taken from all participants. Study will be conducted in 6 weeks' time period. Data will be collected at the start of research and after six week post research date will collected for analysis. Patients will be allocated randomly into two main groups. Group A is the interventional group and group B is the control group. On group A snag will be performed and Group B will be provided by cervical manipulation to compare the effects of both techniques. SPSS will be used for data entry and analysis.

DETAILED DESCRIPTION:
The main aim of the study is to compare the effects of sustained natural apophyseal glides versus cervical manipulation on pain and disability in Nonspecific acute neck pain among wrestlers. Acute neck pain and disabilities are most common among wrestlers. Different studies occur on snags and mobilizations on various athletes but there is a literature gap between comparison of Snags and cervical manipulation in neck disabilities.

This study will be conducted to evaluate effect of sustained natural apophyseal glides and cervical manipulation in pain and disability of neck among wrestler players .All subjects will be selected between ages 18 to 35 years. Data will be collected from players in registered gujranwala wrestling clubs. Study design will be Randomized Clinical Trial. Neck pain disability index questionnaire and NPRS will be used to check the disability in neck and intensity of pain respectively. Informed consent will be taken from all participants. Study will be conducted in 6 weeks' time period. Data will be collected at the start of research and after six week post research date will collected for analysis. Patients will be allocated randomly into two main groups. Group A is the interventional group and group B is the control group. On group A snag will be performed and Group B will be provided by cervical manipulation to compare the effects of both techniques. SPSS will be used for data entry and analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years male only
* Acute non-specific neck pain

Exclusion Criteria:

* Patients with history of discogenic cause in neck.
* History of Postoperative patients
* Individuals who was not willing and individuals with systemic disorders
* Any musculoskeletal(MSK) injury that effect their performance like fracture and bruises etc.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Professional and Elite Male wrestlers of Pakistan
Enrollment: 56 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Numeric pain Rating scale(NPRS) | 6 Weeks
  Pain is rated on single 11 point scale in which 0 indicates no pain and 10 indicates possible worst pain. All individuals will be asked to point out the number mention on the scale. The exact values will be recorded and used for analysis.
NECK DISABILITY INDEX (NDI) | 6 Weeks
  NDI score varies from 0 to 50.Zero is the most desirable state of health.Value 50 is the least desirable state of health.NDI score varies from 0 to 50. Zero is the most desirable state of health.Value 50 is the least desirable state of health.
  Each of the 10 item is scored 0 to 5. The maximum score therefore 50.All the subjects will be asked to circle or tick the one choice from the given sections which most closely describe their problem. The overall item average score will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Durall CJ. Therapeutic exercise for athletes with nonspecific neck pain: a current concepts review. Sports Health. 2012 Jul;4(4):293-301. doi: 10.1177/1941738112446138. PMID 23016100
- [Background] Ali A, Shakil-Ur-Rehman S, Sibtain F. The efficacy of Sustained Natural Apophyseal Glides with and without Isometric Exercise Training in Non-specific Neck Pain. Pak J Med Sci. 2014 Jul;30(4):872-4. PMID 25097535
- [Background] Verhagen AP. Physiotherapy management of neck pain. J Physiother. 2021 Jan;67(1):5-11. doi: 10.1016/j.jphys.2020.12.005. Epub 2020 Dec 24. No abstract available. PMID 33358545
- [Background] Moutzouri M, Billis E, Strimpakos N, Kottika P, Oldham JA. The effects of the Mulligan Sustained Natural Apophyseal Glide (SNAG) mobilisation in the lumbar flexion range of asymptomatic subjects as measured by the Zebris CMS20 3-D motion analysis system. BMC Musculoskelet Disord. 2008 Oct 1;9:131. doi: 10.1186/1471-2474-9-131. PMID 18828921
- [Background] Clark R, Doyle M, Sybrowsky C, Rosenquist R. Epidural steroid injections for the treatment of cervical radiculopathy in elite wrestlers: case series and literature review. Iowa Orthop J. 2012;32:207-14. PMID 23576942